CLINICAL TRIAL: NCT01563484
Title: Comparison of Liver and Renal Function After TACE for PHC With Iso-osmolar and Low-osmolar Contrast Media
Brief Title: Comparison of Liver and Renal Function After Transarterial Chemoembolization for Primary Hepatocellular Carcinoma With Iso-osmolar Contrast Media and Low Osmolar Contrast Media
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Li Chen (Other)
Responsible Party: Sponsor-Investigator, Li Chen, Zhongda Hospital, Southeast University Nanjing, Jiangsu, China, Southeast University, China
Organization: Southeast University, China (Other)
Other Study IDs: 320982198703092517
Record Dates: First submitted 2012-03-20; First posted 2012-03-27 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Primary Hepatocellular Carcinoma
Keywords: Primary Hepatocellular Carcinoma(HCC); Transarterial chemoembolization (TACE); Liver function; Renal function
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- low-osmolar contrast media: Patients undergo TACE of low-osmolar contrast media on day 1.
- iso-osmolar contrast media: Patients undergo TACE of iso-osmolar contrast media on day 1.

SUMMARY:
Primary Hepatocellular Carcinoma (PHC) is one of the most common malignant tumors in the world. In men is the fifth most frequently diagnosed cancer worldwide but the second most frequent cause of cancer death. In women, it is the seventh most commonly diagnosed cancer and the sixth leading cause of cancer death. An estimated 748,300 new liver cancer cases and 695,900 cancer deaths occurred worldwide in 2008. Half of these cases and deaths were estimated to occur in China. Surgical resection and liver transplantation can be curative treatment options, but less than 20% of PHC patients are candidates for surgery. The prognosis of patients with unresectable PHC is poor; if left untreated, the median survival is less than 6 months. Since transarterial chemoembolization (TACE) was introduced as a palliative treatment in patients with unresectable HCC, it has become one of the most common forms of interventional therapy. However, the possibility of treatment-related complication may offset the survival benefit, especially by the worsening of liver functions.TACE increases several parameters of hepatic cytolysis and decreases the metabolic activity of the liver. Such a deterioration of liver function due to ischemia following TACE may result in liver failure, or even death. TACE also may have an adverse effect on the kidney. Radiographic contrast medium is used to obtain the hepatogram before TACE. It has been shown that the use of contrast medium increases the risk of renal failure, especially the low-osmolar contrast media. The aim of this trials was to compare the change of liver and renal function after TACE for HCC of iso-osmolar contrast media with that of low-osmolar contrast media.

DETAILED DESCRIPTION:
This was a prospective, randomized, single centre, single-blind study. Patients were randomized (1:1) to use Low-osmolar contrast media or iso-osmolar contrast media for TACE.

On the morning of 2th and 5th days after TACE, a hematologic check was performed, the hematologic check including serum creatinine, blood urea nitrogen, direct bilirubin, indirect bilirubin, alanine aminotransferase, aspartate aminotransferase, γ-glutamyltransferase, lactate dehydrogenase, alkaline phosphatase, cholinesterase. Then, comparing them with the data before TACE.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years;
* PHC that could not be treated with surgery;
* Patients with clear consciousness，Cooperation;
* Informed consent: authorization and signature.

Exclusion Criteria:

* Preexisting dialysis;
* Known hypersensitivity to the contrast media;
* Complete portal vein thrombosis (main trunk or both branches);
* With severe cardiovascular or renal disease;
* Extensive arteriovenous shunting;
* Insufficient function of the remaining liver (Child-Pugh class C).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This test chooses the patients with unresectable PHC. Then divide them into two groups.In one group,patients underwent a transarterial infusion of ioversol injection(a kind of low-osmolar contrast media).In the other group,patients underwent a transarterial infusion of iodixanol injection(a kind of iso-osmolar contrast media).
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in serum creatinine, blood urea nitrogen, direct bilirubin, indirect bilirubin, alanine aminotransferase, aspartate aminotransferase, γ-glutamyltransferase, lactate dehydrogenase, alkaline phosphatase, cholinesterase. | Follow-up on the 2th and 5th days after TACE

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, MD, Principal Investigator — Medical School,Southeast University
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China